CLINICAL TRIAL: NCT02419820
Title: Randomized, Double-blind, Placebo-controlled, Dose-escalation, Repeated and Single Oral Dosing Phase I Study to Assess the Pharmacokinetics, Pharmacodynamics and Safety of Temanogrel Co-administered With Aspirin and Clopidogrel
Brief Title: Dose-escalation, Repeated and Single Oral Dosing Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Collaborators: Asan Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: ID-TMG-102
Record Dates: First submitted 2015-01-27; First posted 2015-04-17 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — APD791; Clopidogrel; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (16):
- APD791 10mg single dose (Experimental): APD791 10mg single dose
  Interventions: Drug: APD791
- APD791 20mg single dose (Experimental): APD791 20mg single dose
  Interventions: Drug: APD791
- APD791 40mg single dose (Experimental): APD791 40mg single dose
  Interventions: Drug: APD791
- APD791 10mg (Experimental): APD791 10mg single dose + Aspirin + Clopidogrel
  Interventions: Drug: APD791; Drug: Clopidogrel; Drug: Aspirin
- APD791 20mg (Experimental): APD791 20mg single dose + Aspirin + Clopidogrel
  Interventions: Drug: APD791; Drug: Clopidogrel; Drug: Aspirin
- APD791 40mg (Experimental): APD791 40mg single dose + Aspirin + Clopidogrel
  Interventions: Drug: APD791; Drug: Clopidogrel; Drug: Aspirin
- APD791 80mg (Experimental): APD791 80mg single dose + Aspirin + Clopidogrel
  Interventions: Drug: APD791; Drug: Clopidogrel; Drug: Aspirin
- APD791 160mg (Experimental): APD791 160mg single dose + Aspirin + Clopidogrel
  Interventions: Drug: APD791; Drug: Clopidogrel; Drug: Aspirin
- APD791 240mg (Experimental): APD791 240mg single dose + Aspirin + Clopidogrel
  Interventions: Drug: APD791; Drug: Clopidogrel; Drug: Aspirin
- APD791 320mg (Experimental): APD791 320mg single dose + Aspirin + Clopidogrel
  Interventions: Drug: APD791; Drug: Clopidogrel; Drug: Aspirin
- APD791 Placebo (Placebo Comparator): APD791 placebo for single dose + Aspirin + Clopidogrel
  Interventions: Drug: APD791; Drug: Clopidogrel; Drug: Aspirin; Drug: Placebo for APD791
- APD791 2mg MD (Experimental): APD791 2mg multiple dose + Aspirin + Clopidogrel
  Interventions: Drug: APD791; Drug: Clopidogrel; Drug: Aspirin
- APD791 5mg MD (Experimental): APD791 5mg multiple dose + Aspirin + Clopidogrel
  Interventions: Drug: APD791; Drug: Clopidogrel; Drug: Aspirin
- APD791 10mg MD (Experimental): APD791 10mg multiple dose + Aspirin + Clopidogrel
  Interventions: Drug: APD791; Drug: Clopidogrel; Drug: Aspirin
- APD791 20mg MD (Experimental): APD791 placebo for multiple dose + Aspirin + Clopidogrel
  Interventions: Drug: APD791; Drug: Clopidogrel; Drug: Aspirin
- APD791 placebo MD (Placebo Comparator): APD791 placebo for multiple dose + Aspirin + Clopidogrel
  Interventions: Drug: APD791; Drug: Clopidogrel; Drug: Aspirin; Drug: Placebo for APD791

INTERVENTIONS:
Drug: APD791 — Temanogrel
  Other Names: Temanogrel
Drug: Clopidogrel — Clopidogrel
  Other Names: Plavix
  Arms: APD791 10mg; APD791 10mg MD; APD791 160mg; APD791 20mg; APD791 20mg MD; APD791 240mg; APD791 2mg MD; APD791 320mg; APD791 40mg; APD791 5mg MD; APD791 80mg; APD791 Placebo; APD791 placebo MD
Drug: Aspirin — Aspirin
  Other Names: Aspirin Protect
  Arms: APD791 10mg; APD791 10mg MD; APD791 160mg; APD791 20mg; APD791 20mg MD; APD791 240mg; APD791 2mg MD; APD791 320mg; APD791 40mg; APD791 5mg MD; APD791 80mg; APD791 Placebo; APD791 placebo MD
Drug: Placebo for APD791 — Placebo for APD791
  Other Names: Placebo for Temanogrel
  Arms: APD791 Placebo; APD791 placebo MD

SUMMARY:
Randomized, Double-blind, Placebo-controlled, Dose-escalation, Repeated and Single Oral Dosing Phase I Study to Assess the Pharmacokinetics, Pharmacodynamics and Safety of APD791 (Temanogrel) Co-administered with Aspirin and Clopidogrel.

DETAILED DESCRIPTION:
1. To investigate pharmacokinetic and pharmacodynamic characteristics of Temanogrel when orally co-administered with Aspirin and/or Clopidogrel in healthy subject. a person determined to be suitable for the purpose of this clinical trial by investigator with consideration for the age and the health status of a volunteer is selected
2. Assess the safety of Temanogrel when orally co-administered with Aspirin and/or Clopidogrel in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. a healthy adult between 20 and 45 years old at the time of visit for screening
2. a person who is able to give written consent
3. a person between 50 and 85 kg at the time of visit for screening
4. a woman who is negative on a serum hCG test at the time of visit and the day before a trial, and who is not nursing, a woman who agrees on double contraception, medically approved, from the time of visit for screening to 90 days after the last administration of a clinical trial drug, or who had a contraceptive operation no later than 120 days before visit for screening, or who is menopausal, a man who had a contraceptive operation no later than 120 days before visit for screening, or who agrees on double contraception, medically approved, from the time of visit for screening to 90 days after the last administration of a clinical trial drug, and also agree not to donate sperm
5. a person more than hemoglobin 12 g/dL at the time of screening (a woman more than hemoglobin 11 g/dL)
6. a person whose vital signs were in the normal range at the time of visit for screening, or who is medically determined not to be clinically significant by an investigator

Exclusion Criteria:

1. a person with the medical history of gastric ulcer, duodenal ulcer or esophageal ulcer within 90 days from the time of visit for screening
2. a person with the medical history of gastrointestinal diseases(e.g. Crohn's disease, ulcerative colitis, etc.) or surgery(excluding uncomplicated appendectomy or herniotomy) affecting the absorption of a clinical trial drug
3. a person with the medical history of blood coagulation disorder or hemorrhagic diseases, or with clinically significant abnormal findings decided by a investigator on blood coagulation test at the time of screening
4. a woman with the medical history of dysfunctional uterine bleeding within a year from the time of visit for screening
5. a person with the medical history of epilepsy or convulsion
6. a person with the medical history of internal organ transplant
7. a person expected to be hard to complete a clinical trial because of surgery or medical procedures planned within a clinical trial period
8. a person with the medical history of clinically significant new diseases within 30 days from the time of visit for screening according to investigator's decision
9. a person with hypersensitivity reaction to a drug or gelatin, or the medical history of clinically significant hypersensitivity reaction
10. a person with the history of drug abuse, or with a positive reaction to a drug possible to be abused on urine drug screening
11. a person with the medical history of alcohol abuse within two years from the time of visit for screening
12. a person who is a smoker, or with a positive reaction on a urine nicotine test conducted at the time of visit for screening
13. a person who donated whole blood within 60 days or constituents of blood within 30 days, or received a blood transfusion within 30 days from the time of visit for screening
14. a person taking other clinical trial drugs within 90 days from the time of visit for screening
15. a person taking a prescription drug within 30 days, or a contraindicated drug or oriental medicine within 14 days from the time of visit for screening
16. a person with a positive reaction to a serum test(hepatitis B test, hepatitis C test, HIV test, syphilis test)
17. a person with hepatic enzymes(AST, ALT) more than 2.5 times of the reference upper limit(UNL) or total bilirubin more than 1.5 times of the reference upper limit(UNL) or creatinine more than 1.25 times of the reference upper limit(UNL)
18. a person expected to be hard to complete a clinical trial due to physical or mental status according to investigator's medical decision at the time of visit for screening

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics-Cmax | Day1, Day2, Day3, Day4, Day 7
Pharmacokinetics-Tmax | Day1, Day2, Day3, Day4, Day 7
Pharmacodynamics-% inhibition of serotonin-stimulated platelet aggregation | Day1, Day2, Day4, Day7, Day 8
Pharmacodynamics-change of serotonin-stimulated platelet aggregation | Day1, Day4, Day7
Pharmacodynamics-% inhibition of TRAP-induced platelet aggregation | Day1, Day4, Day7 of every dose for mutiple dose group and first day for single dose group.

SECONDARY OUTCOMES:
adverse event monitoring | up to post-study visit(8day±2)
physical examination | up to post-study visit(8day±2)
vital signs | up to post-study visit(8day±2)
ECG | up to post-study visit(8day±2)
laboratory test | up to post-study visit(8day±2)

CONTACTS AND LOCATIONS:
Overall Officials: Gyunseop Bae, M.D., Principal Investigator — Asan Medical Center